CLINICAL TRIAL: NCT02002507
Title: Effect of Different Surgical Positions on the Cerebral Venous Drainage: an Ultrasound Study on Neurosurgical Patients
Brief Title: Jugular Venous Flow Neurosurgical Patients
Status: Withdrawn | Type: Observational
Why Stopped: We faced technical problem before conducting this study
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr., University Health Network, Toronto
Other Study IDs: 13-6432
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Jugular Venous Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- park bench position: Comparing jugular venous flow in supine and park bench position in neurosurgical patients requiring their surgery in park bench position
  Interventions: Other: comparison of different neurosurgical position
- prone position: Comparing the jugular venous flow in the supine and prone position in patients requiring their surgery to be done in the prone position.
  Interventions: Other: comparison of different neurosurgical position

INTERVENTIONS:
Other: comparison of different neurosurgical position — in 2 of 3 positions (supine, plus either prone or park bench) with both left and right internal jugular vein cross-sectional area of vein, doppler velocity, internal jugular venous flow, position of internal jugular vein in relation to carotid artery (All measured with the use of ultrasound)

SUMMARY:
Our hypothesis is that there will be a decrease in internal jugular venous flow in the park bench position when compared to the supine position. There will also be a change in blood flow between the right and left internal jugular veins in the park bench position. In particular, there will be a greater reduction of flow on the dependent side. However, the internal jugular venous flow will be the same in both the prone and supine positions.

DETAILED DESCRIPTION:
The different positions used in neurosurgery for better accessibility to the operating field (park bench, prone) can impact cerebral venous drainage due to the effects of internal jugular venous outflow of blood, and may increase intracranial pressure. Excessive neck flexion and rotation in the park bench position, or flexion in the prone position, may lead to kinking or twisting of the internal jugular vein. This has been hypothesized as the major cause of disturbed venous drainage during surgery and may lead to neck swelling, brachial plexus injury, macroglossia (swollen tongue), delayed airway obstruction, and increases in intracranial pressure in postoperative patients. Optimal brain perfusion is best in the neutral position of the head, but surgery cannot always be performed in this position. Thus, we look to measure the internal jugular venous flow at different positions, as there have been few studies looking at this important contributing factor.

ELIGIBILITY:
Inclusion Criteria:

* Adult neurosurgical patients who are above the age of 18
* Patients undergoing neurosurgery requiring general anesthesia and placement in either in prone or park bench position for surgical accessibility

Exclusion Criteria:

* Lack of informed consent
* Patients undergoing surgical procedures only in the supine position
* Patients needing a central venous catheter in the neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical patients in either park bench or prone position for their surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11-21 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Jugular venous flow | 1 day
  One of the following will be compared depending on the position of the patient
  * Bilateral internal jugular venous flow in supine and prone position
  * Bilateral internal jugular venous flow in supine and park bench position

SECONDARY OUTCOMES:
cross- sectional area of internal jugular vein | 1 day
  Comparing the cross-sectional area of the internal jugular vein in different positions
doppler velocity of jugular venous flow | 1 day
  Comparing the doppler velocity of jugular venous flow in different surgical positions in neurosurgical patients

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, Principal Investigator — University Health Network, Toronto Western Hospital; Vincent Chan, Principal Investigator — University Health Network, Toronto Western Hospital; Pirjo Manninen, Principal Investigator — University Health Network, Toronto Western Hospital; Audrey MY Tan, Principal Investigator — University Health Network, Toronto Western Hospital; Jigesh Mehta, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (1):
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada